



# TRANSPLANTAČNO-NEFROLOGICKÉ ODDELENIE TRANSPLANT-NEPHROLOGY DEPARTMENT

## STUDY TITLE

# **Predicting Outcomes in Diabetes via microRNA**

**PRODIGY** 

**NCT** number:

In Martin, Slovakia 27th May 2025







# TRANSPLANTAČNO-NEFROLOGICKÉ ODDELENIE TRANSPLANT-NEPHROLOGY DEPARTMENT

# 1. Research Question and Objectives:

- Primary Research Question: Can specific microRNA profiles at 3 months post-kidney transplant predict the development of PTDM?
- **Secondary Research Question:** How do traditional risk factors (age, immunosuppression, obesity, CMV infection) and their interaction with specific
- **Primary Objective:** To identify a panel of microRNAs at 3 months post-kidney transplant that are significantly associated with the development of PTDM within a defined follow-up period (e.g., 1 year, 2 years).

# Secondary Objectives:

- To assess the association between traditional risk factors (age, immunosuppression, obesity, CMV infection) and the development of PTDM.
- To investigate the interaction between specific microRNAs and traditional risk factors in predicting PTDM.
- To explore the correlation between specific microRNA expression

### 2. Study Design:

• Type: Prospective Observational Cohort single center Study

## 3. Study Population:

### • Inclusion Criteria:

- Adult patients undergoing kidney transplantation.
- o Absence of pre-existing type 1 or type 2 diabetes mellitus.
- Willingness to provide informed consent and comply with study procedures.

#### • Exclusion Criteria:

- Pre-existing type 1 or type 2 diabetes mellitus.
- o Previous organ transplantation.
- Severe comorbidities that could confound the assessment of PTDM (e.g., pancreatic disease).
- Inability to provide informed consent.

## • Recruitment:

- Consecutive enrollment of eligible patients undergoing kidney transplantation at your center(s).
- Total Sample Size: 64 patients (PTDM group) + 64 patients (non-PTDM group) =
   128 patients

#### 4. Data Collection and Procedures - see table 1:

#### • Baseline Data:

- Demographics (age, sex, ethnicity)
- Medical history (including pre-transplant comorbidities)
- o Transplant-related data (donor source, cold ischemia time, etc.)
- o Immunosuppression regimen (specific drugs and dosages)
- Weight, height (for BMI calculation)
- CMV status (pre- and post-transplant)
- 3-Month Visit:







### TRANSPLANTAČNO-NEFROLOGICKÉ ODDELENIE

#### TRANSPLANT-NEPHROLOGY DEPARTMENT

- Blood sample for microRNA profiling (collect and store appropriately for later analysis)
- Oral Glucose Tolerance Test (oGTT) Follow standardized protocols for administration and interpretation.

#### • 12-month Follow-up:

- Regular monitoring for the development of PTDM (based on established diagnostic criteria, e.g., ADA criteria).
- Collection of data on immunosuppression changes, CMV infections, and other relevant clinical events.
- Define a specific follow-up period (e.g., 1 year, 2 years) to determine the incidence of PTDM.

#### 5. Outcome Measures:

- **Primary Outcome:** Development of PTDM within the defined follow-up period (diagnosed according to ADA criteria or other established criteria).
- Secondary Outcomes:
  - o Specific microRNA expression levels at 3 months.
  - o Correlation between microRNA expression and oGTT results.
  - Association between traditional risk factors and PTDM.
  - Interaction between microRNAs and traditional risk factors in predicting PTDM.

## 6. Data Analysis:

# • Statistical Methods:

- Repeated Measures Analysis: statistical methods that can handle repeated measures data, such as repeated measures ANOVA or mixed-effects models.
- Correlation Analysis: correlation between microRNA expression levels and the results of the standard oGTT







# TRANSPLANTAČNO-NEFROLOGICKÉ ODDELENIE TRANSPLANT-NEPHROLOGY DEPARTMENT

| | base line | M3 | M12 |
|----------------------------------------------------|-----------|----|-----|
| Age at KT (years) | Х | | |
| Donor type (SCD/ECD/living) | Х | | |
| Weight (kg) | Х | Х | Х |
| Waist circumference (cm) | Х | Х | Х |
| BMI (kg/m²) | Х | Х | Х |
| ADPKD (yes/no) | Х | | |
| Duration of dialysis (months) | Х | | |
| Family history of DM* | Х | | |
| Induction (basiliximab/ATG) | Х | | |
| TAC level (ng/ml) | | Х | Х |
| Corticosteroid dose (mg/day) | | Х | Х |
| History of acute rejection | | Х | Х |
| - If yes, treatment (CS/IA/PF/IVIg/Rtx/dara) | | Х | Х |
| OGTT – standard** | Х | Х | Х |
| HbA1c (%) | | Х | Х |
| C-peptide (µg/l) fasting + 2 hours after meal | | Х | Х |
| Immunoreactive insulin (mU/l) + 2 hours after meal | | Х | Х |
| HOMA-IR | | Х | Х |
| eGFR (ml/min) | | Х | Х |
| Creatinine (µmol/l) | | Х | Х |
| cholesterol (mmol/l) | | Х | Х |
| LDL (mmol/l) | | Х | Х |





# TRANSPLANTAČNO-NEFROLOGICKÉ ODDELENIE

## TRANSPLANT-NEPHROLOGY DEPARTMENT

| HDL (mmol/l) | X | Х |
|------------------------|---|---|
| Triglycerides (mmol/l) | X | Х |
| Hb (g/I) | X | Х |
| CMV PCR (cop/ml) | X | Х |
| microRNA | X | |

M – month, KT – kidney transplantation, SCD – donor with standard criteria, ECD – donor with expanded criteria, BMI – body mass index, ADPKD – autosomal dominant polycystic kidney disease, DM – diabetes mellitus, ATG – antithymocyte globulin, TAC – tacrolimus, KS – corticosteroids, IA – immunoadsorption, PF – plasma exchange, IvIg – intravenous immunoglobulins, RTx – rituximab dara – daratumumab, oGTT – oral glucose tolerance test, HbA1c – glycated hemoglobin, eGFR – estimated glomerular filtration rate (according to CKD-EPI), LDL – low-density lipoproteins, HDL – high-density lipoproteins, Hb – hemoglobin, CMV – cytomegalovirus, PCR – polymerase chain reaction

Table 1



<sup>\*</sup>Parents, grandparents, siblings, children

<sup>\*\*</sup> OGTT will be performed in patients without antidiabetic treatment (insulin and/or oral antidiabetics)